CLINICAL TRIAL: NCT00565981
Title: Subcutaneous MabCampath® (Alemtuzumab) and Oral Fludara® (Fludarabinephosphate) for the Treatment of Refractory or Relapsed Chronic Lymphocytic Leukemia in 2nd or 3rd Line of Treatment: A Pilot Trial (FLUSALEM) for the Determination of Safety, Efficacy and Molecular Profiling for the Prediction of Response
Brief Title: A Pilot Trial With Subcutaneous Alemtuzumab and Oral Fludarabinephosphate for the Determination of Safety, Efficacy and Molecular Profiling for the Prediction of Response
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Arbeitsgemeinschaft medikamentoese Tumortherapie (Other)
Collaborators: Schering-Plough (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FLUSALEM
Record Dates: First submitted 2007-11-29; First posted 2007-11-30 (Estimated); Last update posted 2017-12-07 (Actual); Status verified 2017-12

CONDITIONS: B-cell Chronic Lymphocytic Leukemia
Keywords: B-CLL; refractory; molecular profiling; alemtuzumab; fludarabinephosphate
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — fludarabine phosphate; Alemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Overall study (Experimental): The FLUSALEM protocol combines 4 cycles of oral fludarabine phosphate (40mg/m² d1-3; q 29d) and an intensive dose schedule of alemtuzumab (30mg sc.3 times weekly for 16 weeks) in an outpatient setting
  Interventions: Drug: Fludarabine phosphate; Drug: Alemtuzumab

INTERVENTIONS:
Drug: Fludarabine phosphate — orally, 40 mg/m2 d1-3 q4w, x4 cycles
  Other Names: Fludara®
Drug: Alemtuzumab — subcutaneous, starting dose 3 mg and escalation to 10 mg, then 30 mg, followed by 30 mg thrice weekly for 16 weeks in escalated dose
  Other Names: MabCampath®

SUMMARY:
Open label multicenter, two-step, non-randomized (pilot) study to analyze the safety of 4 cycles of 3-day 40mg/m2 oral fludarabine with simultaneous thrice weekly application of 30mg alemtuzumab s.c. in patients with B-CLL disease in 1st and 2nd relapse after any primary treatment or with disease refractory to any therapy in 1st or 2nd line (including Fludarabine, ). This regimen is preceded by an escalation phase with 3-10-30 mg of alemtuzumab s.c.

After the first phase (completed treatment of 7 patients) an interim analysis of safety and efficacy will be performed. In case of a sufficient risk benefit assessment followed by the enrollment of further 21 patients. Final analysis of safety and preliminary efficacy will be based on all patients enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients with CD23+, CD5+, CD19+, light chain monoclonal B CLL
* 1st or 2nd relapse after fludarabine or any other primary treatment regimen or refractory to primary or secondary treatment (including fludarabine) and simultaneously indication for treatment according to the NCI Workshop Criteria 1996
* Age 19-75
* WHO performance score 0-2
* Informed consent given by the patient

Exclusion Criteria:

* HIV positive or positive for Hepatitis B or C
* active uncontrolled infection
* child bearing age without adequate control of fertility, pregnant or lactating women
* intolerance towards any ingredient of either oral fludarabine or alemtuzumab
* allergy against foreign proteins
* previous treatment with alemtuzumab
* treatment with an experimental drug within the previous 2 months
* second malignant disease (non CLL)
* CLL in transformation (Richter syndrome)
* decreased kidney-function with creatinine-clearance < 30ml/min
* severe concomitant diseases or major organ dysfunctions
* patients who are unable to comply with the requirements of the protocol

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2004-03; Primary Completion 2008-02-13 (Actual); Study Completion 2008-02-13 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | within the duration of study
Complete and overall response rate | within the duration of study
Infections grade III, IV | within the duration of study
Rate of CMV reactivation | within the duration of study

SECONDARY OUTCOMES:
Time to retreatment | within duration of trial
Overall survival | within duration of trial
Response in lymphatic compartments | within duration of trial
Molecular response/ immunologic MRD response | within duration of trial
Quality of Life | within duration of trial

CONTACTS AND LOCATIONS:
Overall Officials: Richard Greil, MD, Principal Investigator — IIIrd Medical Department for Hematology, Oncology, Rheumatology, Infectiology and Hemostasiology at the Medical University of Salzburg
Locations (8):
- Austria (8):
  - Landeskrankenhaus Feldkirch, Feldkirch
  - A.ö. Landeskrankenhaus Fürstenfeld, Fürstenfeld
  - Universitätsklinik Innsbruck/ Klinik für Innere Medizin, Innsbruck
  - A.ö. Landeskrankenhaus Leoben, Leoben
  - Krankenhaus der Stadt Linz, Linz
  - St. Johanns LK, Salzburg
  - A.ö. Krankenhaus der Landeshauptstadt St. Pölten, Sankt Pölten
  - Klinikum Kreuzschwestern Wels GmbH, Wels